CLINICAL TRIAL: NCT06523153
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of a SARS-CoV-2-directed Monoclonal Antibody in Healthy Participants
Brief Title: A Study of the Investigational Monoclonal Antibody, VYD2311, in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Invivyd, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: VYD2311-1-001
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- VYD2311 (Experimental): Injection in healthy volunteer
  Interventions: Biological: VYD2311
- Placebo (Placebo Comparator): Injection in healthy volunteer
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VYD2311 — Monoclonal antibody
  Arms: VYD2311
Other: Placebo — Matching Placebo
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
A study to investigate the safety, tolerability, and pharmacokinetics of a SARS-CoV-2-directed monoclonal antibody in healthy participants

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, randomized, double blind, placebo controlled, single escalating dose study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of VYD2311, a monoclonal antibody targeting SARS-CoV-2, in healthy volunteers.

The primary objective is to evaluate the safety and tolerability of multiple dose levels of VYD2311 after a single IV, IM, or SC administration in healthy participants. The secondary objectives are to evaluate the PK of VYD2311 after IV or IM administration and the immunogenicity of VYD2311 after IV, IM, or SC administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female participant aged 18 to 65 years, inclusive.
* Has a body mass index 18.0 to 32.0 kg/m2, inclusive.
* Is in good health, with no clinically significant abnormalities as determined by the Investigator based on medical history, physical exam, vital signs, ECG, and laboratory values per study unit standard operating procedures.
* Tests negative for current SARS-CoV-2 infection by rapid antigen test on screening and Day -1.
* For participants assigned female sex at birth:

  * Is not of childbearing potential (defined in protocol), OR
  * Is of childbearing potential (defined in protocol) and practicing highly effective contraception (defined in protocol) for at least 28 days before dosing (Day 1) through 6 months after dosing and has negative results on pregnancy tests at Screening and on Day -1.
* Is able and willing to provide written informed consent.
* Is able to understand the study procedures and willing to adhere to all protocol requirements.

Exclusion Criteria:

* Has a known or suspected allergy, intolerance, or hypersensitivity to any component of the study drug, including excipients and closely related compounds (eg, other mAbs).
* Intends to receive a COVID-19 vaccine/booster within 3 months of Day 1.
* Is pregnant, breastfeeding, or seeking pregnancy while on study.
* Has any chronic or significant medical condition that, in the assessment of the Investigator, might compromise participant safety or interfere with evaluation of the study drug or interpretation of participant safety/study results, including but not limited to significant neurologic, renal, hepatic, hematologic, immune, cardiac, pulmonary, metabolic, endocrine, psychiatric, vascular, or gastrointestinal disorders.
* Has a history of a malignancy (or active malignancy), except for participants with basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix who have been treated and cured.
* Has had any symptoms of acute respiratory illness (eg, cough, shortness of breath, sore throat, fatigue, loss of smell, fever), or other febrile illness within 2 weeks prior to dosing.
* Has evidence of active infection with HIV, HBV, or HCV, as indicated by any of the following: positive antibody, antigen, or nucleic acid amplification test result for HIV; positive HBV surface antigen; positive HCV antibody with positive HCV RNA (positive antibody test with negative RNA test is not exclusionary).
* Has current alcoholism or recreational drug use, including a positive test result for marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines, or alcohol.
* Is a current or former regular cigarette smoker (more than 5 cigarettes per day within the last year). Individuals who currently or previously smoked 5 or fewer cigarettes per day are allowed if they agree to abstain from smoking during confinement at the CRU.
* Has donated more than 500 mL of blood within 60 days before the scheduled dose of study drug.
* Had major surgery within 30 days prior to study drug dosing or has planned surgeries within 12 months after planned study drug dosing.
* Received any investigational drug or biologic within 30 days or 5 half-lives (whichever is longer) prior to Screening or planned administration of any investigational drug or biologic during the study period.
* Received immunoglobulin or blood products within 6 months prior to Screening
* Previously received a mAb within 6 months or 5 half-lives (whichever is longer) prior to Screening or previously received pemivibart (VYD222) at any time.
* Has taken prescription or OTC medications or supplements within 5 half-lives of the specific substance (or, if half-life is not known, within 48 hours) before the scheduled administration of study drug, with the following exceptions:

  * Influenza or COVID-19 vaccination more than 14 days prior to dosing, or any other vaccine more than 4 weeks prior to dosing
  * Hormonal contraceptives
  * Standard of care use of acetaminophen/paracetamol
  * Vitamins and other nutritional supplements that are not newly introduced (ie, have been taken for at least 30 days prior to enrollment)
  * Other OTC medications that, in the judgement of the Investigator or medically qualified designee, will not impact the safety of the participant or data integrity of the study.
* Screening or predose systolic blood pressure that repeatedly measures below approximately 100 mm Hg. If systolic blood pressure measures below 100 mm Hg, the measurement may be repeated twice. If the average of all three measurements is greater than or equal to 100 mm Hg, the participant may be considered eligible as determined by the Investigator or medically qualified designee.
* In the opinion of the Investigator, is unable to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of TEAEs (including AEs and SAEs) | Through Month-6 visit

SECONDARY OUTCOMES:
PK parameter of VYD2311, AUC0-inf (area under the concentration-time curve from time 0 extrapolated to infinity) | Through Month-6 visit
PK parameter of VYD2311, AUClast (area under the concentration-time curve from time 0 to the last quantifiable concentration) | Through Month-6 visit
PK parameter of VYD2311, AUC0-t (area under the concentration-time curve from time 0 to t) | Through Month-6 visit
PK parameter of VYD2311, Cmax (maximum serum concentration) | Through Month-6 visit
PK parameter of VYD2311, Tmax (time to reach maximum serum concentration) | Through Month-6 visit
PK parameter of VYD2311, CL (clearance) | Through Month-6 visit
PK parameter of VYD2311, t1/2 (half-life) | Through Month-6 visit
PK parameter of VYD2311, Vss (apparent volume of distribution at steady state) | Through Month-6 visit
PK parameter of VYD2311, Vz (apparent volume of distribution during terminal phase) | Through Month-6 visit
Incidence of ADAs against VYD2311 | Through Month-6 visit

CONTACTS AND LOCATIONS:
Locations (1):
- Invivyd Investigative Site, Joondalup, WA 6027, Australia

IPD SHARING:
Plan to Share IPD: No